CLINICAL TRIAL: NCT06143410
Title: Does Intravenous Lidocaine Reduce ED 50 for Propofol Administered Using Target Controlled Infusion (TCI) During Gastroscopy in ASA 1 and 2 Patients.
Brief Title: Intravenous Lidocaine to Reduce ED50 for Propofol Administered Using Target Controlled Infusion (TCI) During Gastroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SRB2023309
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-11

CONDITIONS: Diagnostic Gastroscopy
MeSH Terms: interventions — Lidocaine; Propofol; Gastroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: computered randomisation, sealed enveloppes linisol versus placebo prepared by anesthesist not involved in the study or in patient care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linisol (Active Comparator): Patients will receive 1.5 mg/kg of intravenous linisol before propofol sedatation and gastroscope introduction
  Interventions: Drug: Lidocaine 2% Injectable Solution; Drug: Propofol injection; Procedure: gastroscopy
- Control (Placebo Comparator): Patients will receive intravenous placebo (saline solution),before propofol sedation and gastroscope introduction
  Interventions: Drug: Saline administration as placebo; Drug: Propofol injection; Procedure: gastroscopy

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — administration of a bolus of lidocaine 1.5 mg/kg
  Arms: Linisol
Drug: Saline administration as placebo — administration of a bolus of saline solution as a placebo
  Other Names: administration of a bolus of saline solution as a placebo
  Arms: Control
Drug: Propofol injection — Sedation by total intravenous administration (TIVA) of propofol using target controlled infusion (TCI)
Procedure: gastroscopy — esogastroduodenoscopy

SUMMARY:
The goal of this prospective, interventionnal clinical trial is to assess if intravenous administration of linisol reduce the ED50 of propofol when administered using Target Controlled Infusion (TCI) during gastroscopy in healthy patients (ASA 1 and 2 patients).

Prior to propofol sedation, participants will receive either an intravenous bolus of linisol (1.5 mg/kg) = treated group or placebo = control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for gastroscopy under narcosis and who have signed the consent.
* ASA score: 1 and 2
* BMI between 18 and 30 kg/m2

Exclusion Criteria:

* Lidocaine allergy
* Anesthesia within the last 7 days
* Use of local anesthesia in the last 24 hours
* Rhythm disorder or HR <50
* Pregnant women and breastfeeding
* Participation in another clinical study in the last months
* Cannot understand VAS score or French
* Severe central nervous disease and mental illness.
* Obstructive sleep apnea (known or STOP BANG score >5)
* Upper lung infection.
* Liver or kidney function disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
ED50 of propofol | gastroscope introduction
  ED50 of propofol for gastroscope introduction without movements

SECONDARY OUTCOMES:
number of participants with moderate hypoxemia | Procedure (during propofol sedation and gastroscopy)
  pulse saturation below 95%
number of participants with hypotension | Procedure (during propofol sedation and gastroscopy
  mean arterial pressure below 65 mmHg
number of participants presenting cough | Procedure (during propofol sedation and gastroscopy)
  cough suggesting to light sedation
number of participants presenting laryngospasm | Procedure (during propofol sedation and gastroscopy)
  laryngospasm suggesting to light sedation
number of participants presenting involuntary movements | Procedure (during propofol sedation and gastroscopy)
  involuntary movements suggesting to light sedation
number of participants presenting side effects of lidocaine administration | Time Frame: during gastroscopy procedure
  metallic taste, tinnitus, anaphylaxis
score of Endoscopist satisfaction (1-5) | completed procedure (before transfer to recovery room)
  Endoscopist satisfaction :1 = very bad; 2=bas; 3=good; 4=very good; 5= excellent
score of Patient satisfaction (1-5) | at recovery room discharge, an average of 1 hour after completed procedure
  Patient satisfaction :1 = very bad; 2=bas; 3=good; 4=very good; 5= excellent
throat pain | at recovery room discharge, an average of 1 hour after completed procedure
  analog digital scale from 1 to 10
Time to anesthesia recover | completed procedure (before transfer to recovery room)
  Time between stopping Propofol and recovering a MOAA/S score ≥ 4
Time for post anesthesic care unit discharge | at recovery room discharge, an average of 1 hour after completed procedure
  Time between arrival and discharge of the post anesthesic care unit (Aldrette score >9)

CONTACTS AND LOCATIONS:
Overall Officials: Céline Boudart, PhD, Principal Investigator — Erasme University Hospital
Locations (1):
- Boudart Céline, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after publication
Access Criteria: data will be provided anonymously upon request by email from the corresponding author